CLINICAL TRIAL: NCT06622707
Title: EFFECT OF KINESIO TAPING ON POST-C-SECTION PAIN AND COMFORT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Şırnak Üniversitesi (Other)
Responsible Party: Principal Investigator, Kübra Akcan, lecturer, Şırnak Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 78
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: C-Section
Keywords: Kinesio Taping; Pain; Postpartum Comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesio taping group (Experimental): Kinesio taping will be applied to this group.
  Interventions: Other: kinesio taping; Other: Routine clinical care
- control group (Experimental): Participants in this group will not receive any intervention other than routine clinical care.
  Interventions: Other: Routine clinical care

INTERVENTIONS:
Other: kinesio taping — Despite the increasing indications and new application techniques developed all over the world, it is believed that there is a need for evidence regarding the mechanisms of action and effectiveness of kinesio taping. As a result of the literature review, no study was found in which kinesio taping was applied for 72 hours as a non-pharmacological complementary method to reduce postoperative pain after cesarean section and increase postpartum comfort. In this study, it is planned to apply kinesiotaping for 72 hours after cesarean section.
  Arms: kinesio taping group
Other: Routine clinical care — As routine clinical care; Analgesic treatment protocol applied after cesarean section, postnatal care and discharge services are provided

SUMMARY:
Kinesio taping gently stretches the skin and creates a gap between the dermis and fascia, increasing lymphatic and vascular flow and reducing pain without restricting movement. It is used to provide rehabilitation after surgical operations. This study will be conducted to determine the effect of kinesio taping on the mother's pain and comfort after cesarean section. It is planned to include 60 women who gave birth by cesarean section in the obstetrics and gynecology department at Şırnak State Hospital. Research data will be collected with the visual analog scale and postpartum comfort scale. If the data shows normal distribution, Unrelated Samples t Test, Related Samples t Test and Repeated Measures ANOVA (Repeated Measures) tests will be used.

ELIGIBILITY:
Inclusion Criteria:

* patients having C-section delivery in the 37th and 40th gestational weeks,
* patients giving birth to just a baby,
* patients with no chronic disease (such as allergy, diabetes, or hypertension),
* patients having no problems with communication,
* patients with no dermatological disease.

Exclusion Criteria:

* patients whose babies are in the neonatal intensive care unit,
* patients with deep vein thrombosis, open wounds, or skin irritation,
* patients who did not want to participate in the study,

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who have had a cesarean section will be included in the study.
Enrollment: 60 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
vas | VAS will be applied at the 10th hour, 24th hour, 48th hour and 72nd hour after cesarean section.
  It is used to measure subjectively perceived pain
Postpartum comfort questionnaire | It will be filled in at the 10th and 72th hours after birth.
  It is a scale that can be used appropriately and safely in measuring the postpartum comfort of mothers who have given birth normally or by cesarean section, in meeting the postpartum comfort needs, and in evaluating the outcome as a concrete indicator of the outcome.

IPD SHARING:
Plan to Share IPD: Yes
I accept IPD sharing
Supporting Information: Study Protocol